CLINICAL TRIAL: NCT03958526
Title: Effectiveness of Transcranial Direct Current Stimulation in Chronic Pain Related to Lumbar Spinal Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Enes Efe Is, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LSS tDCS
Record Dates: First submitted 2019-04-01; First posted 2019-05-22 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Lumbar Spinal Stenosis
Keywords: transcranial direct current stimulation; non-invasive brain stimulation; neuromodulation; chronic pain; neurogenic claudication
MeSH Terms: conditions — Spinal Stenosis; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Active stimulation over M1
  Interventions: Device: active tDCS
- Sham (Placebo Comparator): Sham stimulation over M1
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: active tDCS — Patients in active group will receive 10 sessions of anodal tDCS delivered over primary motor cortex (M1) contralateral to the most painful side with a constant current of 2 miliAmpers for 20 minutes.
  Arms: Active
Device: sham tDCS — Same protocol (electrode montage,session duration) will be used for sham stimulation. But the device won't be active for full 20 minutes.
  Arms: Sham

SUMMARY:
Transcranial Direct Current Stimulation (tDCS) is a promising non-invasive brain stimulation technique in chronic pain. There is no study investigating the effectiveness of tDCS in radiating chronic lower extremity pain related to lumbar spinal stenosis (LSS). The aim of this study is to investigate the effects of tDCS on pain, walking capacity, functional status and quality of life in patients with chronic pain related to LSS.

32 patients diagnosed with chronic pain related to LSS will be enrolled in this prospective, randomized, double blind, placebo-controlled study according to inclusion/exclusion criteria. Patients in active group will receive 10 sessions of anodal tDCS delivered over primary motor cortex (M1) with a constant current of 2 miliAmpers for 20 minutes. Patients will be evaluated at baseline, on day 1, 5 and 10 (after the session) and 5 days, 1 month and 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Magnetic resonance imaging evidence of narrowing of the central canal, lateral recess, and/or foramen.
* Persistent leg pain for at least 3 months
* An average pain intensity score (during walking) of at least 4 out of 10 on the Visual Analog Scale at screening and randomisation
* Persistent neurogenic claudication for at least 3 months
* stable pharmacological treatment for pain and sleep disorders for at least 1 month before the study and throughout the trial
* If present, coexisting low back pain intensity should be less than leg pain intensity.

Exclusion Criteria:

* Patients with other neurological or psychiatric disorders including ongoing major depression (Beck Depression Score>14)
* Uncontrolled/unstable endocrinologic, cardiovascular, pulmonary, hematologic, hepatic, renal disease
* Inflammatory diseases, cancer
* Severe hip and/or knee osteoarthritis that affects Treadmill Walking Test
* Absolute/relative contraindications of tDCS (past head trauma resulting with loss of consciousness, epilepsy, past neurosurgical intervention, intracranial hypertension, implanted devices, migraine, chronic-severe headache episodes, a history of side effects with non-invasive brain stimulation techniques, skin diseases, pregnancy)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain as measured by Visual Analog Scale | 12 weeks
  The visual analog scale for pain is a straight line, 10 centimeters (10 cm) in length with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. A higher score indicates greater pain intensity (0 (min)-10 (max)) .
Walking Duration and Distance | 12 weeks
  Patients will be asked to walk on a treadmill at zero angle and a self-selected speed until they have to stop due to symptoms of LSS or until a time limit of 30 minutes has been reached. To start the test, the investigator slowly increases the speed to 1.9 km per hour. The subjects will be then allowed to modify the speed during the test to maintain a pace that is comfortable for them. Subjects will be asked to notify the investigator when they first experience a change in symptoms. Subjects will be also asked to avoid holding the handle bars. Total distance and time, distance and time to onset of symptoms will be measured.

SECONDARY OUTCOMES:
Changes in Functional Status | 12 weeks
  The investigators will use the Modified Oswestry Low Back Pain Disability Questionnaire to assess changes in functional status. The Modified Oswestry Disability Index (MODI) is a validated, 10-point patient-reported outcome questionnaire. Each of the 10 questions is scored from 0 to 5, giving a maximum score of 50. The total score is then converted into a percentage by multiplying it by 2. A higher score indicates worse functional status.
Changes in Quality of Life: Short Form-36 | 12 weeks
  The investigators will use the Short Form-36 to assess changes in quality of life. The SF-36 is a 36-item self-report measure of health-related quality of life. It has eight subscales measuring different domains of health-related quality of life: physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role-emotional (RE), and mental health (MH). The SF-36 also includes a single item that assesses perceived change in health status over the past year. Higher scores on all subscales represent better health and functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Enes Efe Is, MD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Is EE, Aksu S, Karamursel S, Ketenci A, Sindel D. Effectiveness of transcranial direct current stimulation in chronic pain and neurogenic claudication related to lumbar spinal stenosis. Neurol Sci. 2024 Feb;45(2):769-782. doi: 10.1007/s10072-023-07248-z. Epub 2023 Dec 13. PMID 38091212